CLINICAL TRIAL: NCT01607476
Title: Bridging Study of C11 PiB and F18 Flutemetamol Brain PET
Brief Title: Bridging Study of C11 Pittsburgh Compound B (PiB) and F18 Flutemetamol Brain Positron Emission Tomography (PET)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Val Lowe, Consultant - Diagnostic Radiology, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12-000118
Record Dates: First submitted 2012-05-23; First posted 2012-05-30 (Estimated); Results first posted 2016-11-01 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2016-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole; flutemetamol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alzheimer's Disease (Experimental): Subjects who have the clinical diagnosis of probable AD ages 50 and older who have a study partner who is the participant's power of attorney (POA) or legally authorized representative (LAR).
  Interventions include C11 PiB PET/CT and F-18 Flutametamol PET/CT with C11 PiB PET/CT performed first.
  Interventions: Drug: C11 PiB; Drug: F18 Flutametamol
- Cognitive Normal Elderly (Active Comparator): Cognitive Normal subjects who are greater than 60 years of age. Interventions include C11 PiB PET/CT and F-18 Flutametamol PET/CT with C11 PiB PET/CT performed first.
  Interventions: Drug: C11 PiB; Drug: F18 Flutametamol
- Cognitive Normal Young (Active Comparator): Cognitively normal subjects who are between 30-60 years old. Interventions include C11 PiB PET/CT and F-18 Flutametamol PET/CT with C11 PiB PET/CT performed first.
  Interventions: Drug: C11 PiB; Drug: F18 Flutametamol

INTERVENTIONS:
Drug: C11 PiB — One time intravenous administration of 8-22 millicurie (mCi) C11 PiB
  Other Names: C11 PiB PET/CT; C11 Pittsburgh Compound B
Drug: F18 Flutametamol — One time intravenous administration of 3-7 mCi F18 Flutametamol.
  Other Names: F18 Flutametamol PET/CT; Vizamyl

SUMMARY:
The intent of this research protocol is to test the equivalency of two amyloid imaging drugs (C11 Pittsburgh Compound B and F18 Flutemetamol). The investigators hypothesize that there will be no significant difference in the distribution of the agents to areas of amyloid deposition in the brain or to other normal brain structures. Recent data have shown similarity in the distribution of the drugs in subjects with Alzheimer's disease (AD) or mild cognitive impairment (MCI). No comparison data of the two PET drugs in normal subjects has been published. It is important to understand differences in the images and biodistribution from the two drugs in normal subjects as nonspecific accumulation of the drugs in brain structures such as white matter appear to differ slightly and could affect image performance.

DETAILED DESCRIPTION:
Some of the current thinking in regards to the pathophysiology of AD involves the production of amyloid Beta protein (AB) by secretase processing of amyloid precursor protein (APP). While AB is thought to be toxic to neurons its role leading to AD pathogenesis, this is not without debate. In any case, it appears that AB forms amyloid plaques that are largely ubiquitous in AD. Neuronal cell death as a result of the disease is another clear pathophysiologic finding. Because of the importance of these findings in the development of AD, targeted therapies are being investigated to selectively inhibit AB production and/or manipulate amyloid load.

Positron emission tomography (PET) is a molecular imaging modality used to noninvasively measure functional processes of the body. A trace amount of a radiopharmaceutical is injected into a patient and the radiopharmaceutical will be taken up or localized in the body as a function of certain biological processes. The detectors of a PET scanner then measure the radiopharmaceutical distribution externally and the reconstructed PET images should represent the true distribution of the radiopharmaceutical within the body.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 30 years of age or older.
2. Subjects who have the clinical diagnosis of probable AD (30) ages 50 and older who have a study partner who is the participant's power of attorney (POA) or legally authorized representative (LAR), cognitive normal elderly (30) age >60 and cognitive normal young subjects (30) ages 30-60.
3. Normal subjects with Clinical Dementia Rating (CDR) 0-0.5 and AD subjects with CDR of 0.5 or greater.

Exclusion Criteria:

1. Subjects unable to lie down without moving for 30 minutes.
2. Women who are pregnant or who cannot stop breast feeding for 24 hours.
3. Standard safety exclusionary criteria for MRI such as metallic foreign bodies, pacemaker, etc,.
4. Subjects who are too claustrophobic to perform the tests.
5. Subject who have had previous brain irradiation, stroke or brain tumor(s)

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Val Lowe, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
This study was funded by an industrial partner (GE) and discussions with the company about sharing the data will be entertained after first publications.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Mayo Clinic in Minnesota.
Pre-assignment Details: 89 subjects were consented, but 1 subject was a screen failure prior to assignment.
Groups:
- Alzheimer's Disease: Subjects who have the clinical diagnosis of probable Alzheimer's disease (AD) ages 50 and older who have a study partner who is the participant's power of attorney (POA) or legally authorized representative (LAR). Interventions include C11 Pittsburgh Compound B (PiB) PET/CT, F-18 Flutametamol PET/CT.
  C11 PiB: One time intravenous administration of 8-22 millicurie (mCi) C11 PiB
  F18 Flutametamol: One time intravenous administration of 3-7 mCi F18 Flutametamol.
- Cognitive Normal Elderly: Cognitive Normal subjects who are greater than 60 years of age. Interventions include C11 PiB PET/CT, F-18 Flutametamol PET/CT.
  C11 PiB: One time intravenous administration of 8-22 mCi C11 PiB
  F18 Flutametamol: One time intravenous administration of 3-7 mCi F18 Flutametamol.
- Cognitive Normal Young: Cognitively normal subjects who are between 30-60 years old. Interventions include C11 PiB PET/CT, F-18 Flutametamol PET/CT.
  C11 PiB: One time intravenous administration of 8-22 mCi C11 PiB
  F18 Flutametamol: One time intravenous administration of 3-7 mCi F18 Flutametamol.
Period: Overall Study
Arm/Group | Alzheimer's Disease | Cognitive Normal Elderly | Cognitive Normal Young
Started | 25 | 30 | 33
Completed | 24 | 30 | 30
Not Completed | 1 | 0 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Alzheimer's Disease: Subjects who have the clinical diagnosis of probable AD (30) ages 50 and older who have a study partner who is the participant's power of attorney (POA) or legally authorized representative (LAR).
  Interventions include C11 PiB PET/CT, F-18 Flutametamol PET/CT.
  C11 PiB: One time intravenous administration of 8-22 mCi C11 PiB
  F18 Flutametamol: One time intravenous administration of 3-7 mCi F18 Flutametamol.
- Total: Total of all reporting groups
Arm/Group | Alzheimer's Disease | Cognitive Normal Elderly | Cognitive Normal Young | Total
Number analyzed (Participants) | 25 | 30 | 33 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 30 | 33 | 88
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 18 | 49
  Male | 13 | 11 | 15 | 39
Region of Enrollment [Number; unit: participants]
  United States | 25 | 30 | 33 | 86

OUTCOME MEASURES:

1. Primary Outcome: Global Distribution of C11 PiB in the Brain
Description: The imaging analysts use a global atlas of the brain to measure the uptake of the radioactive tracer (or brightness) globally. This global uptake was normalized to the uptake in the cerebellar crus region of the brain to get a global Standard Uptake Value Ratio (SUVR). The cerebral crus (crus cerebri) is the anterior portion of the cerebral peduncle which contains the motor tracts.
  The standard uptake value (SUV) is a way of determining activity in PET imaging. The SUVR is the ratio of SUV from two different regions within the same PET image. For the SUVR, the injected activity, the body weight and the volume to mass conversion factor that are all part of the SUV calculation, cancel.
Time Frame: Approximately one hour after injection of positron emission tomography (PET) drug
Measure: Mean (Standard Deviation); unit: standard uptake value ratio
Arm/Group | Alzheimer's Disease | Cognitive Normal Elderly | Cognitive Normal Young
Number analyzed (Participants) | 24 | 30 | 30
standard uptake value ratio | 2.50 (0.53) | 1.47 (0.28) | 1.23 (0.08)
Statistical Analysis 1: Comparison: Alzheimer's Disease vs Cognitive Normal Elderly; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Alzheimer's Disease vs Cognitive Normal Young; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Cognitive Normal Elderly vs Cognitive Normal Young; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Primary Outcome: Global Distribution of F18 Flutemetamol in the Brain
Description: as for outcome 1
Time Frame: Approximately one hour after injection of positron emission tomography (PET) drug
Measure: Mean (Standard Deviation); unit: standard uptake value ratio
Arm/Group | Alzheimer's Disease | Cognitive Normal Elderly | Cognitive Normal Young
Number analyzed (Participants) | 24 | 30 | 30
standard uptake value ratio | 2.49 (0.49) | 1.59 (0.26) | 1.34 (0.09)
Statistical Analysis 1: Comparison: Alzheimer's Disease vs Cognitive Normal Elderly; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Alzheimer's Disease vs Cognitive Normal Young; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Cognitive Normal Elderly vs Cognitive Normal Young; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Participants were followed for adverse events over the 24 hour period after injection with the study drugs.
Arm/Group | Alzheimer's Disease | Cognitive Normal Elderly | Cognitive Normal Young
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/24 | 4/30 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alzheimer's Disease (N=24) | Cognitive Normal Elderly (N=30) | Cognitive Normal Young (N=30)
Decreased vision (Eye disorders) | 0 (0) | 1 (1) | 1 (1) — Event experienced while subjects were on C-11 PIB, determined to be unrelated to study drug
Hypoglycemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Event experienced while subject on F-18 Flutemetamol, determined to be unrelated to study drug.
Heart palpitations (moderate) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Event experienced while subject on F-18 Flutemetamol, determined to be unrelated to study drug.
Metallic taste (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Event experienced while subject was on F-18 Flutemetamol, determined to be not related to study drug.
Leg cramp (mild) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Event experienced while subject was on F-18 Flutemetamol, determined to be unrelated to study drug.
Dizziness (mild) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Event experienced while subject was on F-18 Flutemetamol, determined to be unrelated to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes